CLINICAL TRIAL: NCT02998463
Title: A Skin-to-Skin Contact (SSC) Facilitating Device Used Within a Mother-Infant Dyad: Exploring Its Acceptability, Usage and Effect on Health Outcomes in the Postnatal Period.
Brief Title: Facilitating Skin-to-Skin Contact In the Postnatal Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham City University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Bailey /Nov /2016 /RC /0640
Record Dates: First submitted 2016-12-14; First posted 2016-12-20 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Breast Feeding; Body Temperature Changes
Keywords: Skin-to-skin; Kangaroo Care; Kangaroo Mother Care
MeSH Terms: conditions — Breast Feeding; Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snuby® users (Experimental): This group receives the Snuby® skin-to-skin facilitating garment to use in the first six weeks following birth with their baby. The use of the Snuby® garment is participant led, and used for as long and as often as they wish in the six week period.
  Interventions: Device: skin-to-skin facilitating garment
- Conventional Care (No Intervention): This group does not receive any intervention, and collects data on the research outcomes when having conventionally facilitated skin-to-skin contact, using a towel, blanket, or clothing as preferred. Skin-to-skin contact frequency and duration is dictated by the participant.

INTERVENTIONS:
Device: skin-to-skin facilitating garment — Fabric garment designed to accommodate term neonates having skin-to-skin contact.
  Other Names: Snuby®
  Arms: Snuby® users

SUMMARY:
This study evaluates the safety and efficacy of a skin-to-skin facilitating garment used by mother-infant dyads. It has three phases including researcher observation, randomised controlled trialing and qualitative midwifery staff perspective. The research will determine the effect a facilitating garment has in comparison to conventionally facilitated skin-to-skin contact, by measuring its effect on the baby's temperature stability, breastfeeding status and weight velocity.

DETAILED DESCRIPTION:
Skin-to-skin contact is used as part of a package of Kangaroo Mother Care across the world. This has been demonstrated to reduce neonatal morbidity, mortality, and inpatient stays for low birth weight and preterm infants (Charpak and Ruiz 2016).

This study examines the effect a facilitating garment, the Snuby® has on neonatal health outcomes associated with skin-to-skin contact, such as neonatal thermoregulation, breastfeeding status, and self-reported mother-infant bonding. It uses a mixed methods approach to address quantitative and qualitative outcomes including participant's perspectives, and measurable health markers.

ELIGIBILITY:
Maternal participants

Inclusion Criteria:

Women, non-binary and transgender participants. Aged 16+ years old. Vaginal birth, including ventouse, forceps and spontaneous vaginal birth. 28+ weeks pregnant. Body Mass Index of 18 to 30 inclusive. Births between 37 and 42 completed weeks of pregnancy. Women without any morbidities that will significantly impair their ability to independently parent their baby.

Women planning to give birth on the labour ward, co-located birth centre, standalone birth centre or at home.

Exclusion Criteria:

Caesarean section births. High dependency Unit patients. Illiterate in English. Multiple pregnancies e.g. twins. Registered child protection concerns. Substance misusing women. Body Mass Index of less than 18 at booking appointment. Body Mass Index of more than 30 at booking appointment. Aged under 16 years old.

Neonatal participants

Inclusion criteria:

Born 37 to 42 completed weeks gestation. Birth weight between 2500g and 4000g . Weight at six weeks of age less than 6000g. Neonates requiring blood glucose prefeed monitoring. From birth to six weeks of age.

Exclusion criteria:

Preterm neonates (less than 37 weeks gestation). Requirement for special or intensive neonatal care. Receiving phototherapy. Receiving intravenous antibiotics. Falling growth velocity of more than 2 centiles. Aged over 6 weeks old.

Midwifery staff participants

Inclusion Criteria:

Working at the National Health Service Trust hosting the research. Working through the Hospital Bank. Registered midwife through the Nursing and Midwifery Council. Working on band 5, 6 or 7. Working within the hospital setting.

Exclusion Criteria:

Midwifery staff working in the community without rotating to the hospital wards.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Abnormal neonatal temperature | Following 30 minutes of skin-to-skin contact, in both Intervention and Control groups.
  Axillary temperature taken by the mother with Eco Temp Basic thermometer. Abnormal: less than 36.5°C or more than 37.5°C.

SECONDARY OUTCOMES:
Breastfeeding Status | Assessed at 3 days post birth, then weekly from day of birth until six weeks postnatal.
  Exclusive breastfeeding, mixed breast and formula feeding, exclusive formula feeding, addition of expressed breastmilk. Includes a comparison to self reported antenatal infant feeding intentions.
Mother Infant bonding | Six weeks post birth
  Maternal participants will self report on their perspectives of skin-to-skin contact, and its role in the relationship bonding process between themselves and their babies.
Neonatal Weight Velocity | At a minimum of 3 intervals, including at birth, ten days, and at six weeks post birth.
  Neonatal weight in grams to ensure suitable for Snuby® garment.
Maternal participant's perspective | Weekly until 6 weeks post birth
  Maternal participants will self-report their views on the garment's ease of use and perceived value. This will be compared to the control group reporting on the same outcomes with conventionally facilitated skin-to-skin contact.
Midwifery participant's perspective | 12 months post birth of the first participating mother-infant dyad.
  Qualitative data collection from midwifery participants, including their perspectives on skin-to-skin contact in the hospital setting, and the perceived value of the Snuby® garment.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McIntyre, DHSci, Principal Investigator — University of Leicester
Locations (2):
- United Kingdom (2):
  - Birmingham City University, Birmingham, West Midlands
  - Sandwell and West Birmingham NHS Trust, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charpak N, Ruiz JG. Latin American Clinical Epidemiology Network Series - Paper 9: The Kangaroo Mother Care Method: from scientific evidence generated in Colombia to worldwide practice. J Clin Epidemiol. 2017 Jun;86:125-128. doi: 10.1016/j.jclinepi.2016.05.019. Epub 2016 Oct 17. PMID 27765653